CLINICAL TRIAL: NCT06520774
Title: A Prospective, Multicenter, Single-Group Target-Value Clinical Trial: Concave Supra-arch Branched Stent-Graft System for Endovascular Treatment of Aortic Arch Diseases
Brief Title: Concave Supra-arch Branched Stent-Graft System for Endovascular Treatment of Aortic Arch Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Collaborators: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P134-01
Record Dates: First submitted 2024-07-07; First posted 2024-07-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Aortic Arch Aneurysm; Penetrating Aortic Ulcer
Keywords: Lifetech; Concave Supra-arch Branched Stent-Graft System; Endovascular Treatment
MeSH Terms: conditions — Aneurysm, Aortic Arch; Penetrating Atherosclerotic Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concave Supra-arch Branched Stent-Graft System (Experimental): Endovascular treatment of patients with Aortic Arch Diseases using Concave Supra-arch Branched Stent-Graft System
  Interventions: Device: Concave Supra-arch Branched Stent-Graft System

INTERVENTIONS:
Device: Concave Supra-arch Branched Stent-Graft System — To evaluate the efficacy and safety of Concave Supra-arch Branched Stent-Graft System for endovascular treatment of Aortic Arch Diseases

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of the Lifetech Concave Supra-arch Branched Stent-Graft System for Endovascular Treatment of Aortic Arch Diseases

DETAILED DESCRIPTION:
The physician must strictly adhere to the clinical study protocol and shall not deviate from or substantially alter it. However, in cases of emergency where there is an immediate risk to the subjects that must be eliminated immediately, a report may be submitted in written form afterward. During the study, any amendments to the clinical study protocol, informed consent documents, requests for deviation, and the resumption of a suspended clinical study must receive written approval from the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are aged 18 to 80 years inclusive；
2. Patients diagnosed with aortic arch aneurysms or penetrating ulcers that require intervention, and for whom the proximal end of the stent needs to be anchored in the Z0 zone;
3. Anatomical criteria, including:

   1. Ascending aorta length is greater than or equal to 50 mm (distance from aortic sinus to anterior edge of innominate artery);
   2. The diameter range of the anchoring area at the proximal end of the main body is between 25-45 mm and the length is greater than or equal to 30 mm;
   3. The diameter of the anchored area of supra-arch branch vessels (innominate artery, left common carotid artery, left subclavian artery) is between 5-18 mm, distal anchorage length is greater than or equal to 15 mm;
   4. Distance between the anterior edge of the innominate artery to the posterior edge of the left subclavian artery is less than or equal to 80 mm;
   5. Have a suitable iliac, femoral, and superior arch arterial access;
4. At least two researchers should assess that the subject is a high-risk patient for surgical treatment or has significant contraindications to surgery. It is recommended to refer to the following criteria: a score of ≥6 in the European System for Cardiac Operative Risk Evaluation (EuroSCORE) scoring system.;
5. Patients who understand the purpose of the study, volunteer to participate and sign the informed consent form, and are willing to complete follow-up visits as required by the protocol.

Exclusion Criteria:

1. Patients either with ruptured or infected aneurysms;
2. Patients with aortic dissection;
3. Patients with general or local infections that may increase the risk of endovascular graft infection;
4. Patients with severe stenosis, calcification, or mural thrombus in the stent anchoring area, which is likely to impede stent-graft adherence or affect stent patency;
5. Previous endovascular intervention involving the aortic arch;
6. Underwent open or endovascular surgery for abdominal aorta within the past 3 months;
7. Patients with a history of stroke within the past 3 months (excluding TIA);
8. Patients with aneurysms involving the distal descending aorta and requiring reconstruction of important visceral branch vessels within the abdomen;
9. Patients with a history of myocardial infarction within the past 3 months;
10. Patients with congestive heart failure - NYHA Class IV;
11. Patients allergic to contrast agents, stent and delivery system materials (such as nitinol, polyester, PTFE, nylon polymer materials);
12. Patients with contraindications to anticoagulant or antiplatelet drugs;
13. Patients unable to tolerate general anesthesia;
14. Patients with abnormal liver and kidney function before surgery (ALT or AST more than 5 times the upper limit of normal; serum creatinine (Cr) >150umol/L);
15. Patients with connective tissue diseases, such as Marfan syndrome, Ehlers-Danlos syndrome, or Behcet's disease;
16. Patients with arteritis;
17. Patients with a life expectancy of less than 1 year;
18. Women who are planning to conceive, pregnant or breastfeeding;
19. Patients deemed by the investigator as unsuitable for endovascular treatment;
20. Patients who have participated in other clinical studies and have not withdrawn or been excluded within the 3 months prior to the screening period of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite endpoints | within 30 days post-surgery
  Composite endpoints refer to the occurrence of any of the following within 30 days post-surgery: all-cause mortality, disabling stroke, or permanent paraplegia.
The clinical treatment success rate within 12 months | pre-discharge (up to 14 days) and 12 months postoperatively
  The 12-month clinical treatment success rate is a composite endpoint that includes immediate technical success after surgery and the absence of the following conditions at 12 months postoperatively: death, displacement of the aortic or branch covered stents on CTA follow-up, Type I or III endoleak, branch stent occlusion, and the need for secondary surgical intervention during the follow-up period.

SECONDARY OUTCOMES:
Immediate technical success rate | Immediate intraoperative
  Immediate technical success refers to the successful delivery of the delivery system to the predetermined position, successful deployment of the system, safe removal of the delivery system from the body, and absence of type I and III endoleaks that require intervention on angiography at the end of the procedure, with all branch stents being patent.
Incidence of increase in the maximum diameter of the aneurysm/depth of ulceration by more than 5 mm at 6 months and 12 months postoperatively. | 6 and 12 months postoperatively
  Increase in the maximum diameter of the aneurysm/depth of ulceration> 5 mm
Incidence rate of Type I/III endoleak at Intraoperative, pre-discharge, 6 and 12 months postoperatively | Intraoperative, pre-discharge（up to 14 days）, 6 and 12 months postoperatively
  A Type I endoleak occurs when there is a gap between the graft and the vessel wall at the "seal zones." This gap allows blood to flow alongside the graft into the aneurysm sac, creating pressure within the sac and increasing the risk of rupture. Type I endoleaks often occur when the aneurysm's anatomy is unsuitable for endovascular aneurysm repair (EVAR) or due to inappropriate device selection. However, vessel dilation over time can also cause this type of endoleak. Immediate attention is typically required because of the high risk of sac enlargement and rupture.
  A Type III endoleak results from a defect or misalignment between the components of the endograft. Similar to a Type I endoleak, a Type III endoleak causes systemic pressure within the aneurysm sac, increasing the risk of rupture. Consequently, Type III endoleaks also necessitate urgent attention.
  The definition of "pre-discharge" is either the discharge date or the 14th postoperative day, whichever occurs first.
Incidence rate of stent graft migration at 6 and 12 months postoperatively | 6 and 12 months postoperatively
  Migration is defined according to reporting standards as a stent graft shift of more than 10 mm relative to a primary anatomic landmark, or any displacement that results in symptoms or necessitates therapy. A standardized measurement protocol was employed in accordance with the reporting guidelines.
The patency rate of the branch vessel at 6 and 12 months postoperatively | 6 and 12 months postoperatively
  Branch vessel patency is defined as stenosis of ≤50%
Incidence rate of secondary surgical interventions related to the aortic arch and its branch arteries before discharge , at the 6 months and 12 months , and at 2-5 years postoperatively | before discharge （up to 14 days）, at the 6 months and 12 months , and at 2-5 years postoperative
  Incidence of secondary surgical interventions related to the aortic arch and its branch arteries
Incidence rate of aneurysm rupture at Intraoperative, pre-discharge, 6 and 12 months, 2-5 years postoperatively | Intraoperative, pre-discharge (up to 14 days）, 6 and 12 months 2-5 years postoperatively
  An aneurysm is an abnormal bulge or ballooning in the wall of a blood vessel. If an aneurysm ruptures, it causes internal bleeding, which can often be fatal.
Incidence rate of delivery system-related complications during perioperative period (from surgery to 30 days after surgery) | perioperative period (from surgery to 30 days after surgery)
  The incidence rate of related complications during the perioperative period (from surgery to 30 days post-surgery) includes intraoperative conversion surgeries due to delivery devices, as well as bleeding, hematoma, and pseudoaneurysm occurring along the delivery access route.
Incidence rate of MAE at Intraoperative, pre-discharge and within 30 days postoperatively | Intraoperative, pre-discharge（up to 14 days） and within 30 days postoperatively
  A Major Adverse Event (MAE) is defined as any occurrence of all-cause mortality, intestinal necrosis, kidney failure, stroke (excluding TIA), permanent paraplegia, myocardial infarction, or respiratory failure.
All-cause mortality at 6 months, 12 months, and 2-5 years postoperatively | 6 months, 12 months, and 2-5 years postoperatively
  All-cause mortality refers to the rate of death from any cause within a specific population over a defined period of time.
Aortic-related mortality at 6 months, 12 months, and 2-5 years postoperatively | 6 months, 12 months, and 2-5 years postoperatively
  Aortic-related mortality refers to the proportion of deaths attributed to aortic conditions within a specific population over a defined period of time.
Incidence rate of severe adverse events at 6 months, 12 months, and 2-5 years postoperatively | 6 months, 12 months, and 2-5 years postoperatively
  A serious adverse event (SAE) in a clinical trial refers to any incident that results in death or a significant deterioration in health. This includes life-threatening illnesses or injuries, permanent impairment of a body structure or function, hospitalization or extended hospital stay, and medical or surgical interventions necessary to prevent permanent damage to physical structure or function. Additionally, SAEs encompass events causing fetal distress, fetal death, or congenital anomalies or defects.
Incidence rate of Device-related adverse events at 6 months, 12 months, and 2-5 years postoperatively | 6 months, 12 months, and 2-5 years postoperatively
  Medical device adverse events are unexpected incidents that occur during or after the use of a medical device by a patient. The World Health Organization (WHO) defines an adverse event as "a problem that can or does result in permanent impairment, injury, or death to the patient or the user." This definition implies two key requirements for determining a medical device adverse event. First, the event must be related to the usage of the medical device. Second, it must be assessed whether the use of the medical device could cause direct harm or potential harm.

CONTACTS AND LOCATIONS:
Overall Officials: chang shu, Professor, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (17):
- China (16):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
  - Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou
  - The First Affiliated Hospital of Kunming Medical University, Kunming
  - The First People's Hospital of Yunnan Province, Kunming
  - Yunnan Fuwai Cardiovascular Disease Hospital, Kunming
  - Jiangsu Provincial People's Hospital, Nanjing
  - Nanjing First Hospital, Nanjing
  - Zhongshan Hospital of Fudan University, Shanghai
  - Shenzhen Hospital of Fuwai Hospital of Chinese Academy of Medical Sciences, Shenzhen
  - Renmin Hospital of Wuhan University, Wuhan
  - Cardiovascular Disease Hospital Affiliated to Xiamen University, Xiamen
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Universitäts-Herzzentrum Freiburg - Bad Krozingen, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No